CLINICAL TRIAL: NCT05994326
Title: Perioperative Care and Short-term Outcomes of Colorectal Surgery: A Prospective Study From Tikur Anbessa Specialized Hospital in Addis Abeba Ethiopia
Brief Title: Perioperative Care and Short-term Outcomes of Colorectal Surgery in Addis Abeba
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Åsa Hallqvist Everhov, Principal investigator, Ass professor, Karolinska Institutet
Other Study IDs: Dnr: 2019-03867
Record Dates: First submitted 2023-07-24; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational cohort study of adult patients undergoing colorectal surgery at Tikur Anbessa Specialized Hospital in Addis Abeba for 3 months.

DETAILED DESCRIPTION:
Observational prospective cohort study, including all adult (≥18) patients undergoing colorectal surgery at Tikur Anbessa Specialized Hospital in Addis Abeba for 3 months. Variables are patients' characteristics, risk factors, investigations, types of operations, level of training of surgeon, and postoperative management. The data collection is conducted at admission, day of surgery, and discharge. The primary outcomes are in-hospital complications and length of stay, and the secondary outcomes are perioperative management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Willingness and ability to give informed consent
* Admitted to the surgical department at TASH (elective or in an emergency) and operated for a colorectal condition

Exclusion Criteria:

-Emergency conditions usually managed in general surgery, e.g., perianal conditions and adhesive small bowel obstruction

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with willingness and ability to give informed consent, who were admitted to the surgical department at TASH (elective or in an emergency) and operated for a colorectal condition
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-12-11 (Actual); Study Completion 2022-12-11 (Actual)

PRIMARY OUTCOMES:
Proportion postoperative complications | From date of surgery to date of discharge from hospital or maximun 30 days postoperatively
  Number and proportion (%) of patients with any postoperative complication according to Clavien-Dindo

SECONDARY OUTCOMES:
Mean length of stay | From admission to date of discharge from hospital, up to 30 days
  Mean number of days in hospital
Type of surgery performed | From admission to date of discharge from hospital, up to 30 days
  Number and proportion (%) of colorectal operations performed (colectomy, rectal resection, stoma without resection)

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Everhov, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Tikur Anbessa Specialized Hospital, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No